CLINICAL TRIAL: NCT03804346
Title: Observational Study to Detect Postoperative Residual Curarization in Infantile Patients
Brief Title: Infantile - Postoperative Residual Curarization - Study
Acronym: I-PORC
Status: Completed | Type: Observational
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Christoph Unterbuchner, Principal Investigator, Dr. med. Christoph Unterbuchner, Staff Anaesthesiologist, University of Regensburg
Other Study IDs: 17-449-101
Record Dates: First submitted 2017-12-01; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Residual Curarization; Neuromuscular Blockade; Neuromuscular Monitoring
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Acceleromyography — At the End of Surgery, shortly before Extubation, the TOF-Ratio is measured by an independent investigator using Acceleromyography.

SUMMARY:
The primary object of this study is, to investigate the current procedure of neuromuscular monitoring at a tertiary academic university medical center.

DETAILED DESCRIPTION:
Residual neuromuscular block is known to be a significant but frequently overlooked complication after the use of neuromuscular blocking agents. Aim of this prospective, observational study is to detect the incidence and severity of residual paralysis at a tertiary academic german university medical center.

Methods:

All infantile patients recieving neuromuscular blocking agents are included over a 12 week observational period. At the end of the operation procedure, directly prior to tracheal extubation a train-of-four ratio was assessed quantitatively by an independet observer using the TOF Watch SX monitor. Data related to patient postoperative outcome were collected in the operating theatre, during the way to the postoperative care unit (PACU) and during the stay in the PACU:

* incidence of residual paralysis
* incidence of aspiration, bronchospasm, laryngospasm, oxygen desaturation, airway obstruction,

ELIGIBILITY:
Inclusion Criteria:

* General aneasthesia with muscle relaxation
* Children between 1 Month to 18 Years
* Endotracheal Intubation due to surgical or diagnostical procedures

Exclusion Criteria:

* older than 18 years
* local aneasthesia
* regional aneasthesia
* larynx mask
* patient comes from ICU
* children who are not planned to be extubated

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All children/youths between 1 Month to 18 years who are undergoing general anaesthesia with muscle relaxation due to surgical or diagnostical procedures.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-23 (Actual); Study Completion 2017-07-23 (Actual)

PRIMARY OUTCOMES:
Residual paralysis | Directly prior to extubation
  Rate of residual paralysis after extubation of the infantile patients measured by acceleromyography.

SECONDARY OUTCOMES:
Airway obstruction | 1, 10, 30, 60 minutes after extubation
  Clinical assessment of the upper airway
Oxygen desaturation | 1, 10, 30, 60 minutes after extubation
  Measurement of the oxygen saturation by pulse oxymetry
Bronchospasm, laryngospasm | 1, 10, 30, 60 minutes after extubation
  Clinical assessment the airway

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Unterbuchner, MD, Principal Investigator — University medical center Regensburg, Department of anaesthesiology
Locations (1):
- University Hospital Regensburg, Regensburg, Bavaria, Germany